CLINICAL TRIAL: NCT03822663
Title: The Influence of Caffeine Supplementation on Discipline-Specific Performance and Training Activities in Combat Sports and Speed-Strength Disciplines
Brief Title: The Influence of Caffeine Supplementation on Specific Performance and Training Activities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Krzysztof Durkalec-Michalski, Principal Investigator, Poznan University of Physical Education
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ULS00007
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Supplementation; Sports
Keywords: Sports nutrition; Caffeine; Physical capacity; Exercise performance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine supplementation (Experimental): Group taking oral CAF (Caffeine) supplementation in a different-dose crossover regimen.
  Interventions: Dietary Supplement: Caffeine supplementation
- Placebo treatment (Placebo Comparator): Group taking oral supplementation with placebo.
  Interventions: Dietary Supplement: Placebo treatment

INTERVENTIONS:
Dietary Supplement: Caffeine supplementation — The experimental procedure for each athlete includes an acute CAF supplementation in a different-dose crossover regimen in order to assess whether the dose affects the actual physical capacity and discipline-specific exercise performance (doses: 3.0-, 6.0- and 9.0 mg/kg of body mass, respectively). CAF (pure pharmaceutical caffeine) will be administered in the dissolved form. On testing days, the supplements will be taken 70 min before physical and exercise capacity test session. Between the CAF and PLA or a PLA and CAF treatments, a minimum 7-day washout period will be introduced.
  Arms: Caffeine supplementation
Dietary Supplement: Placebo treatment — The experimental procedure for each athlete will include PLA supplementation. Placebo will be administered in the dissolved form. On testing days, the PLA will be taken 70 min before physical and exercise capacity test session. Between the PLA and CAF or a CAF and PLA treatments, a minimum 7-day washout period will be introduced.
  Arms: Placebo treatment

SUMMARY:
The purpose of this study is to verify the effect of acute caffeine (CAF) and placebo (PLA) supplementation on physical capacity and discipline-specific exercise performance in athletes, in a randomised, double-blind, placebo-controlled crossover trial.

DETAILED DESCRIPTION:
Caffeine (CAF) is often proposed as an ergogenic agent, especially during high-intensity efforts. CAF supplementation may reduce effort-induced multi-faceted symptoms of fatigue and can improve psychomotor functions (like agility or decision-making processes), which is required during the intermittent high-intensity efforts in combat sports and speed-strength disciplines. Moreover, it is suggested that CAF treatment is associated with increased glycolytic activity during simulated or real training/competition bouts, which results in performance and physical capacity improvement.

However, there are hardly any data on the individual CAF-induced and dose-dependent changes in physical capacity and discipline-specific performance in combat sports and speed-strength disciplines. Therefore, the study aims to examine the effect of acute, different-dose CAF ingestion on physical capacity and discipline-specific performance in combat sports and speed-strength athletes, in a randomized, double-blind, placebo-controlled crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate,
* a current medical clearance to practice sports,
* training experience: at least 2 years,
* minimum of 4 workout sessions (in the discipline covered by the study) a week.

Exclusion Criteria:

* current injury,
* any health-related contraindication,
* declared general feeling of being unwell,
* unwilling to follow the study protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in discipline-specific exercise capacity after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the discipline-specific exercise capacity tests carried out at baseline, and after CAF and PLA supplementation
Changes in caffeine and paraxanthine concencentrations in serum and saliva before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the caffeine and paraxanthine concencentrations (μg/mL), and paraxanthine/caffeine ratio in serum and saliva before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation. Additionally CYP1A2 enzyme activity was assessed by the determination of the mean time-corrected PRX/CAF RATIO in saliva.
Changes in reaction and motor time (Vienna Test System) after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the reaction and motor time (Vienna Test System) (ms) before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in postural stability indices (COP velocity, Vcop) (posturographic platform AccuGaitTM) (after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the postural stability indices (COP velocity, Vcop) (posturographic platform AccuGaitTM) (cm/s) before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in postural stability indices (area 95 percentile, Area95) (posturographic platform AccuGaitTM) after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the postural stability indices (area 95 percentile, Area95) (posturographic platform AccuGaitTM) (cm2) before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation

SECONDARY OUTCOMES:
Changes in sports training / competition activities after discipline-specific exercise tests | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the sports training / competition activities after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in rate of perceived exertion after discipline-specific exercise tests | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the Borg Rating of Perceived Exertion (RPE) scale after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in heart rate during discipline-specific exercise tests | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the Heart Rate during and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Analysis of psychological state before and after caffeine supplementation and placebo | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of psychological state by chosen questionnaires was carried out before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Analysis of macronutrients in diets before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the macronutrients in diets (g) was carried out before the execution of exercise protocols on each research visit
Analysis of body composition (fat-free mass, fat mass) | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of body composition (fat-free mass, fat mass) (kg) was carried out before the execution of exercise protocols on each research visit
Analysis of body composition (total body water) | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of body composition (total body water) (%) was carried out before the execution of exercise protocols on each research visit
Changes in lactate and pyruvate concentrations in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the lactate and pyruvate concentration (mmol/L) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Analysis of gene polymorphisms | Baseline
  Assessment of the chosen gene polymorphisms in saliva carried out at baseline

OTHER OUTCOMES:
Changes in white blood cells and hematological indices (red blood cells, RBC) count in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the leukocytes (neutrophils, monocytes, lymphocytes, neutrophils:lymphocytes ratio) and the hematological indices (red blood cells, RBC)(count/L) count in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in hematological indices (hemoglobin concentration, HGB) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the hematological indices (hemoglobin concentration, HGB) (mmol/L) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in hematological indices (hematocrit, HCT) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the hematological indices (hematocrit, HCT) (L/L) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in hematological indices (mean corpuscular volume, MCV; mean platelet volume, MPV) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the hematological indices (mean corpuscular volume, MCV; mean platelet volume, MPV) (fL) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in hematological indices (mean corpuscular hemoglobin mass, MCH) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the hematological indices (mean corpuscular hemoglobin mass, MCH) (fmol) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in hematological indices (mean corpuscular hemoglobin concentration, MCHC) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the hematological indices (mean corpuscular hemoglobin concentration, MCHC) (mmol/L) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in hematological indices (platelet count, PLT) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the hematological indices (platelet count, PLT) (count x 109/L) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in hematological indices (platelet hematocrit, PCT) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the hematological indices (platelet hematocrit, PCT) (cL/L) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in hematological indices (platelet distribution width, PDW; platelet large cell ratio, PLCR; red blood cells distribution width - coefficient of variation, RDW-C) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the hematological indices (platelet distribution width, PDW; platelet large cell ratio, PLCR; red blood cells distribution width - coefficient of variation, RDW-C) (%) in in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in hematological indices (red blood cells distribution width - standard deviation, RDW-S) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the hematological indices (red blood cells distribution width - standard deviation, RDW-S) (fL) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in nutritional status indices (concentration of urea and magnesium) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the nutritional status indices (concentration of urea and magnesium) (mmol/L) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in nutritional status indices (concentration of glucose, calcium and phosphorans) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the nutritional status indices (concentration of glucose, calcium and phosphorans) (mg/dL) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in muscle damage markers (concentration of creatine) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the muscle damage markers (concentration of creatine) (μmol/L) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation
Changes in muscle damage markers (activity of alanine aminotransferase, aspartate aminotransferase, creatine kinase, lactate dehydrogenase)) in capillary blood before and after caffeine supplementation and placebo treatment | Baseline and during 1 day of acute CAF and PLA supplementation
  Assessment of the muscle damage markers (activity of alanine aminotransferase, aspartate aminotransferase, creatine kinase, lactate dehydrogenase) (U/L) in capillary blood before and after discipline-specific exercise tests carried out at baseline, and after CAF and PLA supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Durkalec-Michalski, PhD, Principal Investigator — Department of Sports Dietetics, Poznan University of Physical Education, Poznan, Poland
Locations (1):
- Department of Sports Dietetics, Poznan University of Physical Education, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Shared data will be exclusively related to the level of recorded indicators, without personal data. The data obtained will be attached to scientific publications, depending on the requirements of the journal.

REFERENCES:
- [Derived] Glowka N, Malik J, Aniola J, Zawieja EE, Chmurzynska A, Durkalec-Michalski K. The effect of caffeine dose on caffeine and paraxanthine changes in serum and saliva and CYP1A2 enzyme activity in athletes: a randomized placebo-controlled crossover trial. Nutr Metab (Lond). 2024 Nov 11;21(1):90. doi: 10.1186/s12986-024-00863-3. PMID 39529054
- [Derived] Durkalec-Michalski K, Nowaczyk PM, Glowka N, Grygiel A. Dose-dependent effect of caffeine supplementation on judo-specific performance and training activity: a randomized placebo-controlled crossover trial. J Int Soc Sports Nutr. 2019 Sep 5;16(1):38. doi: 10.1186/s12970-019-0305-8. PMID 31488190